CLINICAL TRIAL: NCT04185571
Title: Influence of the PEPA Membrane on the Undernutrition Syndrome Inflammation in Chronic Hemodialysis
Acronym: NutriPEPA2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theradial (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THE2010-01
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, prospective, multicenter trial, in two parallel arms
Who Masked: Participant
Masking Description: Patients will be randomized and included in one of the following 2 groups group 1: PEPA membrane / group 2: non-adsorbent synthetic membrane . The randomization will be stratified on the center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEPA membrane (Experimental): PEPA membrane is an adsorbant synthetic copolymer (Poly Ester Poly Arylate)
  Interventions: Device: PEPA
- non adsorbent membrane (No Intervention): Comparison with non adsorbent membrane used in routine

INTERVENTIONS:
Device: PEPA
  Arms: PEPA membrane

SUMMARY:
NutriPEPA2 is a randomized, single-blind, prospective, multicenter trial, in two parallel arms to confirm that the adsorbent PEPA membrane may decrease mortality related to inflammation and malnutrition encountered in HD or HDF-treated stage 5 renal failure compared to a non-adsorbent synthetic membrane.

DETAILED DESCRIPTION:
The objective of NutriPEPA2 study is to demonstrate that the use of an adsorbent membrane (PEPA-Poly Ester Poly Arylate synthetic co-polymer membrane) decreases undernutrition (often associated with inflammation) and consequently morbidity, comparing one year mortality in patients with Chronic Kidney Disease (CKD), with severe Protein-Energy Wasting (PEW), treated with dialysis using a non-adsorbent synthetic membrane (Polysulfone or Polyethersulfone) versus an adsorbent membrane (PEPA).

ELIGIBILITY:
Inclusion Criteria:

* Patient with Chronic Renal Insufficiency Stage 5, treated by fistula or permanent catheters,
* Medium albumin (on 3 recent assays) of less than 35 g / l (this assay being carried out by a non-electrophoretic technique),
* PINI score greater than or equal to 1,
* Beginning of the treatment of extra-renal purification by hemodialysis for at least 3 months on a non-adsorbing synthetic membrane (of the Polysulfone, Polyethersulfone, PolyArylethersulfone type) of surface at least equal to that of the PEPA dialyser

Exclusion Criteria:

* Patients allergic to PEPA,
* Patients with insufficient vascular access,
* Patients with digestive syndromes: Hepatopathy, gastrointestinal amyloidosis, chronic diarrhea, myeloma and dysglobulinaemia, neoplasia and hematopathy, a serious illness that is life-threatening in the short term,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2011-07-12 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Possible decrease mortality in patients arm treated with PEPA membrane | one year
  Superiority of mortality with other non-adsorbent membrane versus adsorbent

SECONDARY OUTCOMES:
Evolution of adipocytokines concentration | one year
  Evolution of four types of adipocytokines (ghrelin, leptin, adiponectin, resistin)

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD HORY, Doctor, Principal Investigator — Centre de Néphrologie, 4 ter rue de la Forêt, Avignon, FRANCE
Locations (12):
- France (11):
  - Ch Annonay, Annonay
  - Ch Besancon, Besançon
  - Ch Chartres, Chartres
  - Ch La Rochelle, La Rochelle
  - CH MEAUX, Meaux
  - Ch Metz-Thionville, Metz
  - Aura Paris Plaisance, Paris
  - CH Saint Brieuc, Saint-Brieuc
  - CH Saint Quentin, Saint-Quentin
  - Ch Toulouse Larrey, Toulouse
  - Chru Tours, Tours
- CHPM Monaco, Monaco, MC, Monaco

IPD SHARING:
Plan to Share IPD: No